CLINICAL TRIAL: NCT01673126
Title: Transcranial Direct Current Stimulation in Patients With Disorders of Consciousness: a Sham-controlled Randomised Double Blind Study
Brief Title: Transcranial Direct Current Stimulation in Patients With Disorders of Consciousness
Acronym: tDCS in DOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Aurore Thibaut, Principal Investigator, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009/201
Record Dates: First submitted 2012-08-14; First posted 2012-08-27 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Vegetative State; Minimally Conscious State; Disorders of Consciousness
Keywords: vegetative state; minimally conscious state; disorders of consciousness; transcranial direct current stimulation
MeSH Terms: conditions — Persistent Vegetative State; Consciousness Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anodal tDCS (Active Comparator): Patients received anodal tDCS (on DLPF cortex) during 20 minutes preceded and followed by a clinical assessment (Coma Recovery Scale-Revised)
  Interventions: Device: Anodal tDCS
- sham tDCS (Sham Comparator): Patient received a sham tDCS (5sec of stimulation). The device runs during 20minutes and the anode was placed over the DLPF cortex. A behavioral assessment preceded and followed the stimulation.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: Anodal tDCS — patients received anodal tDCS (on PFDL cortex) during 20 minutes preceded and followed by a behavioral assessment (Coma Recovery Scale Revised)
  Arms: Anodal tDCS
Device: sham tDCS — Patient received a sham tDCS (5sec of stimulation). The device runs during 20minutes and the anode was placed over the DLPF cortex. A behavioral assessment preceded and followed the stimulation.
  Arms: sham tDCS

SUMMARY:
Previous studies showed that anodal transcranial direct current stimulation (tDCS) applied to the left dorsolateral prefrontal (DLPF) cortex transiently improves performance of memory and attention. Investigator assessed the effects of left DLPF-tDCS on Coma Recovery Scale-Revised (CRS-R) scores in severely brain damaged patients with disorders of consciousness in a double-blind sham-controlled experimental design.

DETAILED DESCRIPTION:
Following severe brain damage and coma, some patients may remain in a vegetative state (VS) or minimally conscious state (MCS). At present, there are no evidence-based guidelines regarding the treatment of patients with disorders of consciousness (DOC).

Investigator aim to assess the effect of single session anodal (i.e., excitatory) transcranial direct current stimulation (tDCS) of the left dorsolateral prefrontal cortex (DLPF) on the level of consciousness in DOC patients in a double blind randomized sham controlled study.

tDCS is a form of safe non-invasive cortical stimulation, modulating cortical excitability at stimulation sites via weak polarizing currents, previously reported to transiently improve working memory and attention by stimulating the left DLPF in healthy subjects and patients with stroke, Parkinson's or Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* post-comatose patients
* patients in vegetative/unresponsive or minimally conscious state
* patients with stable cardiorespiratory parameters
* patients free of sedative drugs and Na+ or Ca++ channel blockers (e.g., carbamazepine) or NMDA receptor antagonists (e.g., dextromethorphan)

Exclusion Criteria:

* premorbit neurology antecedent
* patients in coma or <1week after the acute brain insult
* patients with a metallic cerebral implant or a pacemaker (in line with the safety criteria for tDCS in humans)

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Laureys, MD, PhD, Study Chair — Coma Science Group, Cyclotron Research Centre, University and University Hospital of Liège
Locations (1):
- University Hospital of Liège, Liège, Liège, Belgium

REFERENCES:
- [Background] Multi-Society Task Force on PVS. Medical aspects of the persistent vegetative state (1). N Engl J Med. 1994 May 26;330(21):1499-508. doi: 10.1056/NEJM199405263302107. PMID 7818633
- [Background] Giacino JT, Ashwal S, Childs N, Cranford R, Jennett B, Katz DI, Kelly JP, Rosenberg JH, Whyte J, Zafonte RD, Zasler ND. The minimally conscious state: definition and diagnostic criteria. Neurology. 2002 Feb 12;58(3):349-53. doi: 10.1212/wnl.58.3.349. PMID 11839831
- [Background] Nitsche MA, Fricke K, Henschke U, Schlitterlau A, Liebetanz D, Lang N, Henning S, Tergau F, Paulus W. Pharmacological modulation of cortical excitability shifts induced by transcranial direct current stimulation in humans. J Physiol. 2003 Nov 15;553(Pt 1):293-301. doi: 10.1113/jphysiol.2003.049916. Epub 2003 Aug 29. PMID 12949224
- [Background] Nitsche MA, Liebetanz D, Lang N, Antal A, Tergau F, Paulus W. Safety criteria for transcranial direct current stimulation (tDCS) in humans. Clin Neurophysiol. 2003 Nov;114(11):2220-2; author reply 2222-3. doi: 10.1016/s1388-2457(03)00235-9. No abstract available. PMID 14580622
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] Kang EK, Kim DY, Paik NJ. Transcranial direct current stimulation of the left prefrontal cortex improves attention in patients with traumatic brain injury: a pilot study. J Rehabil Med. 2012 Apr;44(4):346-50. doi: 10.2340/16501977-0947. PMID 22434324
- [Background] Boggio PS, Ferrucci R, Rigonatti SP, Covre P, Nitsche M, Pascual-Leone A, Fregni F. Effects of transcranial direct current stimulation on working memory in patients with Parkinson's disease. J Neurol Sci. 2006 Nov 1;249(1):31-8. doi: 10.1016/j.jns.2006.05.062. Epub 2006 Jul 14. PMID 16843494
- [Background] Ferrucci R, Mameli F, Guidi I, Mrakic-Sposta S, Vergari M, Marceglia S, Cogiamanian F, Barbieri S, Scarpini E, Priori A. Transcranial direct current stimulation improves recognition memory in Alzheimer disease. Neurology. 2008 Aug 12;71(7):493-8. doi: 10.1212/01.wnl.0000317060.43722.a3. Epub 2008 Jun 4. PMID 18525028

RESULTS

PARTICIPANT FLOW:
Groups:
- Anodal tDCS: Anodal tDCS (on DLPF cortex) first, hen 2 days of washout, then sham tDCS.
- Sham tDCS: Sham tDCS during first, then 2 days of washout, then anodal tDCS.
Period: Overall Study
Arm/Group | Anodal tDCS | Sham tDCS
Started | 36 (First stimulation (20 minutes) Washout (2 days) Second stimulation (20 minutes)) | 26 (First stimulation (20 minutes) Washout (2days) Second stimulation (20 minutes))
Completed | 32 | 23
Not Completed | 4 | 3
Not completed — change of diagnosis | 4 | 3

BASELINE CHARACTERISTICS:
Population: 36 patients received first the anodal stimulation and 26 received first the sham stimulation.
  Each patient received both stimulation exept for 7 patients. They were excluded due to diagnosis change between the 2 stimulations.
Groups:
- Anodal tDCS First: Patients received anodal tDCS during 20 minutes. Then, washout of 2days. Then sham tDCS.
- Sham tDCS First: Patients received sham tDCS during 20 minutes. Then, washout of 2days. Then andoal tDCS.
- Total: Total of all reporting groups
Arm/Group | Anodal tDCS First | Sham tDCS First | Total
Number analyzed (Participants) | 32 | 23 | 55
Age, Customized [Mean (Standard Deviation); unit: years] | 46 (17) | 40 (19) | 43 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 23 | 16 | 39
Region of Enrollment [Number; unit: participants]
  Belgium | 32 | 23 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change in CRS-R Total Scores
Description: At the group level, assess the modification of CRS-R total scores in anodal tDCS as compared to sham stimulation in VS/UWS and MCS populations
  The Coma Recovery Scale Revised (CRS-R) is a behavioral scale performed at the patient's bedside. It consists of 23 hierarchically arranged items that comprise 6 subscales addressing auditory, visual, motor, verbal, communication, and arousal functions.
  Scoring is based on the presence or absence of specific behavioral responses to sensory stimuli administered in a standardized manner. Maximum scores of each subscale are summed to obtain the total score (from 0 to 23).
  The lowest item on each subscale represents reflexive activity, whereas the highest items represent cognitively mediated behaviors.
Time Frame: Baseline and directly after the tDCS (20 minutes)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Anodal tDCS First: Patients received anodal tDCS first during 20 minutes preceded and followed by a clinical assessment (Coma Recovery Scale-Revised).
  Then, a washout period (2days). Then sham tDCS during 20 minutes preceded and followed by a clinical assessment (Coma Recovery Scale-Revised).
- Sham tDCS First: Patients received sham tDCS first during 20 minutes preceded and followed by a clinical assessment (Coma Recovery Scale-Revised).
  Then, a washout period (2days). Then anodal tDCS during 20 minutes preceded and followed by a clinical assessment (Coma Recovery Scale-Revised).
Arm/Group | Anodal tDCS First | Sham tDCS First
Number analyzed (Participants) | 55 | 55
units on a scale | 12.17 (4.32) | 10.60 (4.19)

2. Secondary Outcome: Influence of Diagnosis on the Results
Time Frame: participants will be followed for the duration of 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Influence of Etiology on the Results
Time Frame: participants will be followed for the duration of 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Influence of Time Since Insult on the Results
Time Frame: participants will be followed for the duration of 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the first stimulation to one month after the end of the 2 stimulations.
Description: We use the GOSE (Glasgow outcome scale extended) to assess a possible decrease (or inscrease) in patient status.
Arm/Group | Anodal tDCS | Sham tDCS
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No